CLINICAL TRIAL: NCT02551159
Title: A Phase III Randomized, Open-label, Multi-center, Global Study of MEDI4736 Alone or in Combination With Tremelimumab Versus Standard of Care in the Treatment of First-line Recurrent or Metastatic Squamous Cell Head and Neck Cancer Patients
Brief Title: Phase III Open Label Study of MEDI 4736 With/Without Tremelimumab Versus Standard of Care (SOC) in Recurrent/Metastatic Head and Neck Cancer
Acronym: KESTREL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419LC00001
Record Dates: First submitted 2015-09-09; First posted 2015-09-16 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: programmed cell death ligand 1 (PD-L1), MEDI4736, Cytotoxic T-lymphocyte-associated antigen 4 {CTLA-4}, PFS, SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; tremelimumab; Cetuximab; Fluorouracil; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy (Experimental): MEDI4736 monotherapy.
  Interventions: Biological: MEDI4736
- Combination Therapy (Experimental): MEDI4736+Tremelimumab combination therapy
  Interventions: Biological: Tremelimumab; Biological: MEDI4736+Tremelimumab
- Standard of Care (Active Comparator): Standard of Care treatment
  Interventions: Biological: Cetuximab; Drug: 5-fluorouracil (5FU); Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: MEDI4736 — Anti-PD-L1 antibody
  Arms: Monotherapy
Biological: Tremelimumab — Anti-CTLA-4 Antibody
  Arms: Combination Therapy
Biological: MEDI4736+Tremelimumab
  Arms: Combination Therapy
Biological: Cetuximab — Monoclonal Antibody
  Arms: Standard of Care
Drug: 5-fluorouracil (5FU) — Chemotherapy Agent
  Arms: Standard of Care
Drug: Cisplatin — Chemotherapy agent
  Arms: Standard of Care
Drug: Carboplatin — Chemotherapy Agent
  Arms: Standard of Care

SUMMARY:
This is a randomized, open-label, multi-center, 3-arm, global Phase III study to determine the efficacy and safety of MEDI4736 + tremelimumab combination or MEDI4736 monotherapy versus SoC (EXTREME regimen) in the treatment of patients with SCCHN who have not received prior systemic chemotherapy for recurrent or metastatic disease.

DETAILED DESCRIPTION:
Patients will be randomized in a 2:1:1 ratio to MEDI4736 + tremelimumab combination therapy, MEDI4736 monotherapy, or SoC. Patients in all arms will continue therapy until progression. Tumor assessments will be performed on computed tomography scans or magnetic resonance imaging scans, preferably with intravenous (IV) contrast. Efficacy for all patients will be assessed by objective tumor assessments every 6 weeks for the first 24 weeks, then every 8 weeks thereafter until treatment discontinuation due to progression or toxicity. All patients will be followed every 3 months for survival after progression is confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of screening
2. Documented evidence of recurrent or metastatic SCCHN (oral cavity, oropharynx, hypopharynx, or larynx).
3. A fresh tumor biopsy for the purpose of screening or an available archival tumor sample. Tumor lesions used for fresh biopsies should not be the same lesions used as RECIST target lesions, unless there are no other lesions suitable for biopsy.
4. No prior systemic chemotherapy for recurrent or metastatic disease
5. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
6. No prior exposure to immune-mediated therapy,

Exclusion Criteria:

1. Histologically or cytologically confirmed head and neck cancer of any other primary anatomic location in the head and neck not specified in the inclusion criteria including patients with SCCHN of unknown primary or non-squamous histologies (eg, nasopharynx or salivary gland)
2. Tumor progression or recurrence within 6 months of last dose of platinum therapy in the primary treatment setting
3. Receipt of any radiotherapy or hormonal therapy for cancer treatment within 30 days prior to first dose of study treatment
4. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Olsson, Study Director; Tanguy Seiwert, Principal Investigator — The University of Chicago, 5841 S Maryland Ave, Chicago, IL 60637
Locations (167):
- United States (17):
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Morristown, New Jersey
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Namur
- Brazil (10):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Ijuí
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (10):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (10):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Mainz
  - Research Site, Tübingen
  - Research Site, Würzburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- India (6):
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Gūrgaon
  - Research Site, Karamsad
  - Research Site, Madurai
  - Research Site, Pune
- Italy (9):
  - Research Site, Cona
  - Research Site, Florence
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Salerno
  - Research Site, Siena
  - Research Site, Torino
- Japan (19):
  - Research Site, Akashi-shi
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kanazawa
  - Research Site, Kitaadachi-gun
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Natori-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Toyoake-shi
  - Research Site, Yokohama
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Las Piñas
  - Research Site, Quezon City
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Research Site, Suceava, Romania
- Russia (9):
  - Research Site, Arkhangelsk
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Ufa
  - Research Site, Yekaterinburg
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Košice
- South Korea (7):
  - Research Site, Cheongju-si
  - Research Site, Hwasun-gun
  - Research Site, Incheon
  - Research Site, Seogu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Jaén
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Marbella
  - Research Site, Málaga
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Pathum Thani
- Ukraine (10):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kapitanivka Village
  - Research Site, Kharkiv Region
  - Research Site, Kirovohrad
  - Research Site, Kryvyi Rih
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Vinnytsia
- United Kingdom (6):
  - Research Site, Bebington
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton
  - Research Site, Taunton
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Seiwert TY, Wildsmith S, Fayette J, Harrington K, Gillison M, Ahn MJ, Takahashi S, Weiss J, Machiels JP, Baxi S, Baker V, Evans B, Morsli N, Jill Walker, Real K, L'Hernault A, Psyrri A. Outcomes in biomarker-selected subgroups from the KESTREL study of durvalumab and tremelimumab in recurrent or metastatic head and neck squamous cell carcinoma. Cancer Immunol Immunother. 2024 Mar 2;73(4):70. doi: 10.1007/s00262-024-03643-3. PMID 38430375
- [Derived] Hwang M, Seiwert TY. Are taxanes the future for head and neck cancer? Pragmatism in the immunotherapy era. Lancet Oncol. 2021 Apr;22(4):413-415. doi: 10.1016/S1470-2045(21)00121-2. Epub 2021 Mar 5. No abstract available. PMID 33684371
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419LC00001&attachmentIdentifier=b4025180-dfd4-4783-a723-cba099a5d9fb&fileName=D419LC00001_-_Protocol_v12__-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419LC00001&attachmentIdentifier=0a933c97-43c4-4fdc-8e9f-af78f3808b67&fileName=D419LC00001_-_SAP_v7,0_-_redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419LC00001&attachmentIdentifier=da78c143-9577-4556-a890-e24f765e4d5f&fileName=D419LC00001_-_CSR_Synposis_-_28Apr2021-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting all the eligibility criteria were randomized 2:1:1 to durvalumab plus tremelimumab combination therapy, durvalumab monotherapy or standard of care.
Groups:
- Durvalumab + Tremelimumab: tremelimumab (75 mg) via IV infusion every 4 weeks for a maximum of 4 doses, and durvalumab (1500 mg) via IV infusion every 4 weeks until disease progression
- Durvalumab: durvalumab (1500 mg) via IV infusion every 4 weeks until disease progression
- Standard of Care (SOC): either cisplatin (at a dose of 100 mg/m2 of body surface area as an IV infusion) or carboplatin (at an area under the concentration curve of 5 mg/mL/min as an IV infusion) on Day 1 of up to six 3-week cycles, and an infusion of 5-fluorouracil (5FU) (at a dose of 1000 mg/m2/day on Days 1 through 4) every 3 weeks, along with 400 mg/m2 of cetuximab on Cycle 1 Day 1 and 250 mg/m2 weekly for up to 6 cycles and maintenance cetuximab at 250 mg/m2 administered via IV infusion weekly thereafter in patients who achieved stable disease (SD) or better upon completion of chemotherapy until disease progression, toxicity, or withdrawal of consent
Period: Overall Study
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Started | 413 | 204 | 206
Full Analysis Set (All patients randomized) | 413 | 204 | 206
Safety Analysis Set (All patients who received at least one dose of study treatment) | 408 | 202 | 196
PD-L1 TC/IC High Subgroup Analysis Set (Patients in the full analysis set with PD-L1 high) | 190 | 99 | 94
Completed | 0 | 0 | 0
Not Completed | 413 | 204 | 206
Not completed — Death | 352 | 174 | 161
Not completed — Withdrawal by Subject | 8 | 5 | 16
Not completed — Patients alive or lost to follow-up at DCO | 53 | 25 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC) | Total
Number analyzed (Participants) | 413 | 204 | 206 | 823
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.56) | 60.2 (10.41) | 60.9 (9.45) | 60.5 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 29 | 32 | 134
  Male | 340 | 175 | 174 | 689
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 298 | 145 | 160 | 603
  Black or African American | 5 | 3 | 2 | 10
  Asian | 109 | 54 | 42 | 205
  Other | 0 | 2 | 2 | 4
  Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Status in the PD-L1 TC/IC High Subgroup - Durvalumab Versus Standard of Care (SOC)
Description: Number of participants with Overall Survival (OS)
Time Frame: From date of randomization until time of final analysis, an average of approximately 4 years
Population: PD-L1 TC/IC subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 190 | 99 | 94
Participants
  Death | 162 | 84 | 77
  Voluntary Discontinuation by subject | 1 | 1 | 3
  Alive or lost to follow up | 27 | 14 | 14
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SOC); Statistical analysis of number of deaths; Test type: Superiority; p = 0.787, Log Rank — 2 sided; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.69 to 1.32]

2. Primary Outcome: Overall Survival (OS) Median Duration in the PD-L1 TC/IC High Subgroup
Description: Time from the date of randomization until death due to any cause (i.e., date of death or censoring - date of randomization + 1)
Time Frame: From date of randomization until time of final analysis, an average of approximately 4 years
Population: PD-L1 TC/IC subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 190 | 99 | 94
Months | 11.2 [9.5 to 13.9] | 10.9 [9.0 to 14.3] | 10.9 [8.3 to 13.4]

3. Secondary Outcome: Overall Survival (OS) Status in the PD-L1 TC/IC High Subgroup - Durvalumab + Tremelimumab Versus Standard of Care (SOC)
Description: Number of participants with Overall Survival (OS)
Time Frame: From date of randomization until time of final analysis, an average of approximately 4 years
Population: PD-L1 TC/IC subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 190 | 99 | 94
Participants | 162 | 84 | 77
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SOC); Test type: Superiority; p = 0.634, Log Rank — 2 sided; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.80 to 1.39]

4. Secondary Outcome: Percentage of Patients Alive at 12, 18 and 24 Months in the PD-L1 TC/IC High Subgroup
Description: Percentage of patients alive
Time Frame: 12, 18 and 24 months after randomization
Population: PD-L1 TC/IC subgroup
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 190 | 99 | 94
% of participants
  at 12 months | 49.3 [42.0 to 56.2] | 48.0 [37.8 to 57.4] | 44.0 [33.6 to 53.8]
  at 18 months | 31.8 [25.3 to 38.5] | 34.7 [25.5 to 44.1] | 30.8 [21.6 to 40.4]
  at 24 months | 23.9 [18.0 to 30.1] | 27.6 [19.2 to 36.6] | 26.4 [17.8 to 35.7]

5. Secondary Outcome: Progression Free Survival (PFS) in the PD-L1 TC/IC High Subgroup
Description: Time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression). Progression is defined using Response Evaluation Criteria in Solid Tumours criteria (RECIST v1.1), as ≥20% increase in the sum of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for the first 24 weeks relative to the date of randomization and then every 8 weeks thereafter, up to approximately 4 years
Population: PD-L1 TC/IC subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 190 | 99 | 94
Months | 2.8 [2.6 to 3.3] | 2.8 [1.7 to 4.2] | 5.3 [4.3 to 5.8]
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SOC); Test type: Superiority; p = 0.287, Log Rank — 2 sided; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.94 to 1.80]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SOC); Test type: Superiority; p = 0.028, Log Rank — 2 sided; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.99 to 1.76]

6. Secondary Outcome: Objective Response Rate (ORR) in the PD-L1 TC/IC High Subgroup
Description: Number (%) of patients with at least 1 visit response of complete response (CR) or partial response (PR). Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) for target lesions (TL) and assessed by MRI or CT: CR: Disappearance of all TLs since baseline; PR: >= 30% decrease in the sum of diameters of TLs; Overall Response (OR = CR + PR)
Time Frame: as for outcome 5
Population: PD-L1 TC/IC subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 190 | 99 | 94
Participants
  Response | 48 | 16 | 47
  No response | 142 | 83 | 47
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SOC); Statistical analysis of number with a response; Test type: Superiority; p < 0.001, Regression, Logistic — 2 sided; Odds Ratio (OR) = 0.19, 95% CI 2-sided [0.10 to 0.37]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SOC); Statistical analysis of number with a response; Test type: Superiority; p < 0.001, Regression, Logistic — 2 sided; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.20 to 0.57]

7. Secondary Outcome: Duration of Response (DoR) in the PD-L1 TC/IC High Subgroup
Description: Time from the date of first documented response until the first date of documented progression or death in the absence of disease progression
Time Frame: as for outcome 5
Population: PD-L1 TC/IC subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 48 | 16 | 47
Months | 6.5 [4.5 to 16.1] | 12.3 [5.6 to NA] — The upper confidence limit was not calculable because of an insufficient number of participants with events. | 4.2 [3.0 to 5.7]

8. Secondary Outcome: Overall Survival (OS) Status in the All-comers (Full Analysis Set)
Description: Number of participants with Overall Survival (OS)
Time Frame: From date of randomization until time of final analysis, an average of approximately 4 years
Population: All-comers (Full analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 413 | 204 | 206
Participants
  Death | 356 | 176 | 171
  Voluntary Discontinuation by subject | 4 | 3 | 6
  Alive or lost to follow up | 53 | 25 | 29
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SOC); Statistical analysis of number of deaths; Test type: Superiority; p = 0.811, Log Rank — 2 sided; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.83 to 1.27]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SOC); Statistical analysis of number of deaths; Test type: Superiority; p = 0.624, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.87 to 1.25]

9. Secondary Outcome: Overall Survival (OS) Median Duration in the All-comers (Full Analysis Set)
Description: as for outcome 2
Time Frame: From date of randomization until time of final analysis, an average of approximately 4 years
Population: All-comers (Full analysis set)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 413 | 204 | 206
Months | 10.7 [9.6 to 12.2] | 9.9 [8.9 to 11.9] | 10.3 [9.0 to 12.1]

10. Secondary Outcome: Percentage of Patients Alive at 12, 18 and 24 Months in the All-comers (Full Analysis Set)
Description: Percentage of patients alive
Time Frame: 12, 18 and 24 months after randomization
Population: All-comers (Full analysis set)
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 413 | 204 | 206
% of participants
  at 12 months | 46.5 [41.6 to 51.2] | 42.8 [35.9 to 49.5] | 43.8 [36.8 to 50.5]
  at 18 months | 30.7 [26.3 to 35.2] | 31.2 [24.9 to 37.7] | 29.7 [23.5 to 36.1]
  at 24 months | 22.9 [18.9 to 27.0] | 24.7 [18.9 to 30.8] | 23.2 [17.6 to 29.2]

11. Secondary Outcome: Progression Free Survival (PFS) in the All-comers (Full Analysis Set)
Description: as for outcome 5
Time Frame: as for outcome 5
Population: All-comers (Full analysis set)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 413 | 204 | 206
Months | 2.8 [2.6 to 2.9] | 2.8 [2.0 to 2.8] | 5.4 [4.4 to 5.7]
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SOC); Test type: Superiority; p = 0.006, Log Rank — 2 sided; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [1.10 to 1.68]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SOC); Test type: Superiority; p = 0.008, Log Rank — 2 sided; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [1.06 to 1.53]

12. Secondary Outcome: Objective Response Rate (ORR) in the All-comers (Full Analysis Set)
Description: as for outcome 6
Time Frame: as for outcome 5
Population: All-comers (Full analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 413 | 204 | 206
Participants
  Response | 90 | 35 | 101
  No response | 323 | 169 | 105
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SOC); Test type: Superiority; p < 0.001, Regression, Logistic — 2 sided; Odds Ratio (OR) = 0.21, 95% CI 2-sided [0.13 to 0.33]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SOC); Test type: Superiority; p < 0.001, Regression, Logistic — 2 sided; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.20 to 0.41]

13. Secondary Outcome: Duration of Response (DoR) in the All-comers (Full Analysis Set)
Description: as for outcome 7
Time Frame: as for outcome 5
Population: All-comers (Full analysis set)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
Number analyzed (Participants) | 90 | 35 | 101
Months | 9.2 [6.0 to 19.6] | 11.9 [4.6 to 17.8] | 4.2 [3.7 to 4.5]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events will be collected from the time of signature of informed consent throughout the treatment period and including the follow-up period (up to 90 days after the last dose of investigational product or until initiation of another therapy) for an average of approximately 4 years.
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 356/413 | 176/204 | 171/206
Serious Adverse Events (participants affected / at risk) | 168/408 | 78/202 | 94/196
Other Adverse Events (participants affected / at risk) | 317/408 | 153/202 | 182/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Tremelimumab (N=408) | Durvalumab (N=202) | Standard of Care (SOC) (N=196)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (14) | 2 (2) | 4 (4)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 4 (4) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 4 (5)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Troponin t increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 1 (1) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 8 (9)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (6)
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 1 (1) | 5 (5)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (12) | 1 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (3) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 3 (3) | 2 (2)
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 3 (3) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 32 (33) | 14 (14) | 13 (13)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 2 (3)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 1 (1) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (2)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Tremelimumab (N=408) | Durvalumab (N=202) | Standard of Care (SOC) (N=196)
Anaemia (Blood and lymphatic system disorders) | 61 (68) | 22 (26) | 65 (97)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 26 (48)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 63 (103)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (24) | 0 (0) | 39 (76)
Hyperthyroidism (Endocrine disorders) | 23 (30) | 6 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 68 (79) | 21 (23) | 7 (7)
Constipation (Gastrointestinal disorders) | 59 (72) | 24 (25) | 54 (68)
Diarrhoea (Gastrointestinal disorders) | 70 (113) | 15 (20) | 60 (96)
Dysphagia (Gastrointestinal disorders) | 26 (28) | 8 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 52 (65) | 13 (14) | 74 (120)
Stomatitis (Gastrointestinal disorders) | 14 (16) | 6 (6) | 40 (54)
Vomiting (Gastrointestinal disorders) | 34 (52) | 8 (9) | 39 (66)
Asthenia (General disorders) | 52 (60) | 18 (23) | 38 (61)
Fatigue (General disorders) | 66 (74) | 35 (41) | 56 (68)
Mucosal inflammation (General disorders) | 15 (16) | 6 (8) | 43 (58)
Pyrexia (General disorders) | 48 (54) | 12 (13) | 21 (33)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 21 (24)
Pneumonia (Infections and infestations) | 19 (22) | 7 (7) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 27 (37) | 8 (10) | 11 (14)
Lipase increased (Investigations) | 21 (27) | 5 (8) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 24 (36)
Platelet count decreased (Investigations) | 5 (5) | 1 (1) | 22 (47)
Weight decreased (Investigations) | 39 (42) | 13 (15) | 26 (32)
Decreased appetite (Metabolism and nutrition disorders) | 52 (57) | 20 (22) | 46 (59)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 16 (27)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (11) | 3 (6) | 45 (77)
Hyponatraemia (Metabolism and nutrition disorders) | 26 (30) | 2 (4) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (27) | 8 (8) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 10 (10)
Dizziness (Nervous system disorders) | 15 (18) | 7 (7) | 14 (15)
Insomnia (Psychiatric disorders) | 29 (31) | 8 (9) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (47) | 14 (14) | 13 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (40) | 5 (5) | 18 (21)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 12 (12) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 11 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 36 (50)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (24) | 4 (4) | 26 (34)
Pruritus (Skin and subcutaneous tissue disorders) | 45 (61) | 11 (13) | 17 (18)
Rash (Skin and subcutaneous tissue disorders) | 50 (62) | 17 (17) | 81 (114)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 18 (23)
Hypertension (Vascular disorders) | 27 (36) | 9 (10) | 11 (19)
Hypotension (Vascular disorders) | 11 (15) | 5 (5) | 11 (16)
Alanine aminotransferase increased (Investigations) | 23 (26) | 6 (6) | 14 (18)
Blood creatinine increased (Investigations) | 15 (20) | 3 (4) | 12 (19)
Dehydration (Metabolism and nutrition disorders) | 8 (10) | 0 (0) | 10 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 29 (37) | 6 (8) | 8 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (26) | 6 (8) | 22 (42)
Headache (Nervous system disorders) | 29 (35) | 11 (12) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02551159/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT02551159/SAP_001.pdf